CLINICAL TRIAL: NCT04436848
Title: Identifying Leucocyte and Urine Biomarkers in Parkinson's Patients With LRRK2 G2385R Gene Variant
Brief Title: LRRK2 G2385R Leucocyte and Urine Biomarker Study
Acronym: LRRK2 G2385R
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); University of Dundee (Other); Nextcea, Inc (Unknown); Max Planck Institute of Biochemistry (Unknown)
Responsible Party: Sponsor
Other Study IDs: UMG2385R
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for extraction of DNA, monocytes and serum Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PD patients positive for LRRK2 G2385R
  Interventions: Other: This is a non-interventional study
- PD patients negative for LRRK2 G2385R
  Interventions: Other: This is a non-interventional study
- Non-PD controls negative for LRRK2 G2385R
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study

SUMMARY:
Given the emerging evidence on LRRK2-related biomarkers, this project will focus on identifying leucocyte and urine biomarkers that are altered by the LRRK2 G2385R variant, and investigating the effects of LRRK2 kinase inhibitor (MLi-2) on these biomarkers, using immunoblotting and mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease assigned by a movement disorder specialist according to clinical diagnostic criteria
* Age above 18 year-old
* Provision of a written informed consent

Exclusion Criteria:

- Physical or mental incapacity to complete study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease attending the Neurology outpatient clinic, at University of Malaya Medical Centre, Kuala Lumpur, Malaysia.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of monocyte-based biomarkers for LRRK2 G2385R variant | Two years
Identification of urine-based biomarkers for LRRK2 G2385R variant | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ai Huey Tan, MD, FRCP, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data will be kept for storage at a central repository either hosted by the funder (Michael J. Fox Foundation), its collaborators, or consultants and will be made publicly available (with no personal identifying information) for the intended use of research in Parkinson's disease as well as other biomedical research studies that may not be related to Parkinson's disease.